CLINICAL TRIAL: NCT05153447
Title: A Multicomponent Technology Supported Care Delivery for Older Patients With Hematologic Malignancies (The M-Tech Study)
Acronym: M-Tech
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain funding
Sponsor: Kah Poh Loh (Other)
Responsible Party: Sponsor-Investigator, Kah Poh Loh, Assistant Professor, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS21086
Record Dates: First submitted 2021-11-16; First posted 2021-12-10 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: Mobile Health Technology; Geriatrics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-Tech (Experimental): M-Tech involves the use of a mobile app delivery platform to several interventions. The components of M-Tech include: 1) Hybrid in-person and telehealth visits with oncology providers; 2) Disease-specific education videos; 3) Activity level monitoring via a wearable device with promotion of physical activity; 4) Symptom monitoring with provision of self-management strategies, and 5) Medication management.
  Interventions: Behavioral: M-Tech
- Usual Care (Active Comparator): Participants randomized to the usual care arm will receive standard of care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: M-Tech — M-Tech involves the use of a mobile app delivery platform to several interventions. The components of M-Tech include: 1) Hybrid in-person and telehealth visits with oncology providers; 2) Disease-specific education videos; 3) Activity level monitoring via a wearable device with promotion of physical activity; 4) Symptom monitoring with provision of self-management strategies, and 5) Medication management.
  Arms: M-Tech
Other: Usual Care — Participants randomized to the usual care arm will receive standard of care.
  Arms: Usual Care

SUMMARY:
This is a randomized controlled trial to assess the feasibility and preliminary efficacy of a multicomponent technology-supported care delivery intervention trial in 110 older patients with hematologic malignancies [acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), multiple myeloma (MM), and diffuse large b-cell lymphoma (DLBCL)] receiving outpatient chemotherapy on treatment-related toxicities, patient-reported outcomes, healthcare utilization, and inflammatory and epigenetic markers.

DETAILED DESCRIPTION:
Compared to younger adults, older adults with cancer are more likely to have age-related vulnerabilities such as functional impairment and co-existing medical conditions. They are also often on many medications. As a result, older adults are more likely to experience treatment-related toxicities. These toxicities can lead to increased healthcare utilization (e.g., hospitalization, emergency room visits), decreased quality of life and functional status, and reduced survival. In addition, a disproportionate number of older adults live in rural areas which often limit access to healthcare. Therefore, there is a need to better support older adults with hematologic malignancies during the course of their treatment to decrease treatment-related toxicities so they can continue to receive treatment. The proposed study will investigate whether digital health technologies can support older adults in various aspects of their cancer care.

ELIGIBILITY:
Inclusion Criteria

* Age ≥60 years
* Have a new diagnosis of AML, MDS, MM, and DLBCL
* Have a plan to receive outpatient chemotherapy for at least 4 months (patients may enroll within the first 2 weeks of chemotherapy initiation if they do not have grade 2 or higher non-hematologic adverse event)
* No plan to or unlikely to proceed with autologous or allogeneic hematopoietic stem cell transplantation (SCT) in the following 5 months (if SCT is planned after 4 cycles of chemotherapy in the case of MDS or myeloma, patients are allowed to enroll)
* English speaking
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* No medical contraindications for exercise per oncologist
* Able to walk 4 meters as part of Short Physical Performance Battery measured walk (with or without the assistive device)
* Able to provide informed consent

Exclusion Criteria:

• None

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between experimental and active comparator arms - Clinician-rated non-hematologic treatment-related toxicity | 4-5 months
  Measured using the Common Terminology Criteria for Adverse Events or CTCAE v5.0 and operationalized based on proportion of patients with grade 3-5 non-hematologic treatment-related toxicity for AML, MDS, and DLBCL or grade 2-5 non-hematologic treatment-related toxicity for MM
Retention rates | 4-5 months
  Percentage of patients/caregivers who completed baseline assessments and subsequently completed post-intervention assessments

SECONDARY OUTCOMES:
Difference between experimental and active comparator arms - Healthcare Utilization | 4-5 months
  Healthcare utilization such as hospitalization and emergency room visits in the first 4-5 months will be collected from medical chart review. These will be presented as proportions and count.
Difference between experimental and active comparator arms - Quality of Life | 4-5 months
  Quality of life, measured using the Functional Assessment of Cancer Therapy-Leukemia (FACT-G) scale. It consists of 27 items divided into 4 subscales: physical well-being (PWB), social well-being (SWB), emotional well-being (EWB), and functional well-being (FWB). The score for each item ranges from 0-4. After reversing the scoring of negatively worded items, all the scores are summated. A higher score indicates better quality of life.
Difference between experimental and active comparator arms - Patient-reported treatment-related toxicity | 4-5 months
  Patient-reported treatment-related toxicity as measured using the Patient-Reported Outcomes version of the CTCAE (PRO-CTCAE). We selected 22 symptoms commonly experienced by older adults with hematologic malignancies. Questions ask about frequency, severity, and interference with daily activities (each question has 5 response options). We will convert these response options to 0-5 and sum up the scores, higher score indicates worse severity and interference.
Difference between experimental and active comparator arms - Functional Status | 4-5 months
  Functional status, measured using the instrumental activities of daily living subscale of the Multidimensional Functional Assessment Questionnaire: Older American Resources and Services (OARS). The IADL subscale consists of seven questions rated on a three-point Likert scale. It measures the degree to which an activity can be performed independently. A higher score indicates better functional status

OTHER OUTCOMES:
Difference between experimental and active comparator arms -Inflammatory cytokines | 4-5 months
  Inflammatory cytokines including TNFα, sTNFR1, sTNFR2, IL-1β, IL-2, IL-6, sIL-6R, IL-8, IL-10 in pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No